CLINICAL TRIAL: NCT02438449
Title: A Cost-Effectiveness Analysis Comparing Abdominal-based Autogenous Tissue (AAT) and Tissue Expander- Implant (TE/I) Reconstruction of the Breast After Mastectomy- A Feasibility Study
Brief Title: Cost-Effectiveness of Abdominal-based Autogenous Tissue vs Tissue Expander-Implant Reconstruction - A Feasibility Study
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Principal Investigator, Achilleas Thoma, Dr. Achilleas Thoma, McMaster University
Other Study IDs: MSA-2015-04
Record Dates: First submitted 2015-04-23; First posted 2015-05-08 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; mastectomy; health-related quality of life; Health Utilities Index; HUI; prospective; quality-adjusted life years; QALY
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Abdominal-based Autogenous Tissue (AAT): The AAT-based breast reconstruction surgery will include any of the following techniques: pedicled transverse rectus abdominis myocutaneous (TRAM) flap, Free TRAM, muscle-sparting TRAM flap, deep inferior epigastric perforator (DIEP) flap, superficial inferior epigastric artery (SIEA) flap, and Rubens flap.
  Interventions: Procedure: Breast Reconstruction Surgery
- Tissue Expander-Implants (TE/I): The TE/I approach will include two-stage breast reconstruction surgery. In the initial stage, immediately after mastectomy and with or without sentinel node biopsy, an expander will be placed in the subpectoral plane and the defect closed. Two weeks after the surgery, the expansion of the TE will commence until the desired volume of the respective expander is achieved. The second stage will include removal of the TE and the placement of a permanent implant which may be either saline or gel. The delayed method will be similar to the immediate reconstruction with the exception of the incision, which will be relatively smaller as the mastectomy was performed previously with breast cavity being fully closed.
  Interventions: Procedure: Breast Reconstruction Surgery

INTERVENTIONS:
Procedure: Breast Reconstruction Surgery — AAT-based orTE/I reconstruction in all patients undergoing breast reconstruction following mastectomy

SUMMARY:
It is estimated that about 25% and 40% of health care expenditures in Canada and USA respectively are wasted because of inefficiencies and not practicing evidence-based medicine. As health care resources are scarce it behooves all of us to use these in a cost-effective manner. The term "cost-effective" is used in the health care literature often but erroneously. Investigators compare a "novel' intervention to a "prevailing" one and if the novel intervention is less costly it is labeled "cost-effective". In a methodologically correct cost-effectiveness study however, investigators need to integrate both the effectiveness and costs of the competing interventions and calculate an incremental cost-effective ratio. If this ratio falls within acceptability thresholds, the novel intervention is labeled cost-effective. There are many techniques of breast reconstruction. The two most common approaches are the Autologous Abdominal Tissue (AAT) and the Tissue Expansion / Implant reconstructions. In this study these two most common breast reconstruction approaches after mastectomy due to cancer performed in the Hamilton/Niagara/Haldimand/Brant and Waterloo/Wellington LHINs will be investigated with a cost-effectiveness analysis coupled with a methodologically robust observational study.

DETAILED DESCRIPTION:
As a result of the recent advances in the treatment of breast cancer carried out by dedicated researchers and made possible through breast cancer research, its mortality has been gradually declining. Naturally, the quality of survivorship has taken an important role in the last 3 decades. Unfortunately, for most women with breast cancer, their concerns about survival are followed closely with concerns about body image, sexuality, self-esteem and social life. Mastectomy, a mainstay in the treatment of breast cancer, is the primary cause of these latter concerns. The investigators are therefore charged with looking at the disease and the respective treatment of breast cancer holistically. Providing a comprehensive management of breast cancer today requires attention to both oncologic principles and to the patient's quality of life. A large part of the patient's quality of life comes from improved reconstructive and aesthetic outcomes following mastectomy. In short, breast reconstruction after mastectomy for cancer aims to improve body image and quality of life by reducing the negative psychological impact of the deformity. Multiple techniques exist to accomplish this goal. They include breast implants, autologous tissues, or occasionally, a combination thereof. Although the ultimate goal is to recreate an aesthetically pleasing breast that attempts to match the missing one, the decision to use a particular technique is multi-factorial. It may be influenced by the surgeon's skills, the patient's preferences, inherent contraindications with a patient, or the resources available in a particular setting. Breast reconstructions can be costly to patients (indirect costs), third party payers and society, especially as new technologies are introduced in clinical practice. In the last 2 decades third party payers and governments in different jurisdictions have been advocating for production of evidence that shows "value for money" germane to these different procedures.Presently, the two most common approaches to breast reconstruction are the AAT method and the TE/I method. These two approaches to breast reconstruction have yet to be submitted to an economic evaluation using state-of-the-art cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Patients undergoing breast reconstruction (immediate or delayed) after mastectomy procedure on one or both breasts.
3. Eligible for two step tissue expander and implant based procedure, or one of the following autogenous abdomen tissue-based procedures (pedicled TRAM flap, Free TRAM, ms TRAM flap, DIEP flap, SIEA flap, Rubens flap).

Exclusion Criteria:

1. Patients who have had previous breast reconstruction surgery.
2. Patients undergoing other procedures during reconstruction surgery, other than the mastectomy itself in the case of immediate or delayed reconstruction.
3. Patients unable to complete the questionnaires due to language barriers.
4. Geographic inaccessibility or inability to adhere to study protocol requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include patients undergoing breast reconstruction after mastectomy on one or both breasts being seen by one of the participating plastic surgeons. If patients qualify for the trial according to the inclusion and exclusion criteria, they will be invited to participate in the study and will be required to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09-01 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life (utilities and disease-specific) | 1 year

SECONDARY OUTCOMES:
Healthcare resource utilization including out-of-pocket expenses by patients | 1 year
  Identify and tabulate the costs for the two procedures under the purview of the patient, Ministry of Health and society. Costs will be further classified into two categories: surgery-related costs and costs incurred by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD MSc FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare / McMaster University, Hamilton, Ontario, Canada